CLINICAL TRIAL: NCT05487781
Title: Phase 1 Clinical Study To Describe the Biological Safety and Pharmacokinetics of Tyrphostin AG-17 Present in Oral Solid Formulations of the Fixed Dose Combination, in Three Different Concentrations of the Compound Tyrphostin AG-17 Content 10 mg, 3.3 mg and 1 mg Respectively, With 700 mg of L-Carnitine Tartrate Each Presentation, in a Single Dose in Healthy Research Subjects of Mexican Nationality
Brief Title: Phase 1 Clinical Study to Describe Biological Safety and Pharmacokinetics of Tyrphostin
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Molecule X LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: F1-TIR-036/0821
Record Dates: First submitted 2022-03-01; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Healthy
Keywords: Phase 1 clinical study; Tirfostin; L-Carnitine; Biological Safety; Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: Assess the biological safety and pharmacokinetics of tyrphostin AG-17 present in the solid oral formulations of the fixed-dose combination, in three different concentrations of the compound tyrphostin AG-17 contained 10 mg, 3.3 mg and 1 mg, respectively, with 700 mg of L-Carnitine tartrate each presentation, in a single dose in healthy research subjects of Mexican nationality.
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator) The random assignment codes to the administration sequence will be under the protection of the Statistics Department. The Analytical Unit, the group of researchers from the Clinical Unit (medical staff) and the IS will remain blinded during the conduct of the study, the processing and analysis of the biological samples and in this way avoid biasing the results generated. Once the Clinical Phase is over, the opening code for the issuance of the Clinical Report and the Safety Report will be shared with the group of researchers of the Clinical Unit (medical staff).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Tyrphostin AG-17 content 10 mg with 700 mg of L-Carnitine tartrate
  Interventions: Combination Product: Tirfostina/L-Carnitina
- Group 2 (Experimental): Tyrphostin AG-17 content 3.3 mg with 700 mg of L-Carnitine tartrate
  Interventions: Combination Product: Tirfostina/L-Carnitina
- Group 3 (Experimental): Tyrphostin AG-17 content 1 mg with 700 mg of L-Carnitine tartrate
  Interventions: Combination Product: Tirfostina/L-Carnitina

INTERVENTIONS:
Combination Product: Tirfostina/L-Carnitina — Estudio clínico fase 1 para describir la seguridad biológica y la farmacocinética de la tirfostina AG-17

SUMMARY:
Evaluate the biological safety and pharmacokinetics of tyrphostin AG-17 present in the solid oral formulations of the fixed-dose combination, in three different concentrations of the compound tyrphostin AG-17 contained 10 mg, 3.3 mg and 1 mg, respectively, with 700 mg of L-Carnitine tartrate each presentation, in a single dose in healthy research subjects of Mexican nationality.

DETAILED DESCRIPTION:
Describe the tolerance of the fixed-dose combination, in three different concentrations of the compound tyrphostin AG-17, containing 10 mg, 3.3 mg and 1 mg, respectively, with 700 mg of L-Carnitine tartrate each presentation, in a single dose in research subjects. healthy Mexican nationals, describing: type, frequency, duration, consequence, relationship with clinical history, management, follow-up; criteria: seriousness, severity; and classification of the AE or ADRs in accordance with the current NOM-220-SSA1 and estimate if there are differences by gender.

Assess the effects on body functions of the fixed dose combination, in three different concentrations of the compound tyrphostin AG-17 content 10 mg, 3.3 mg and 1 mg respectively, with 700 mg of L-Carnitine tartrate each presentation, in a single dose in healthy research subjects of Mexican nationality through the measurement of physiological markers and estimate if there are differences by gender.

Obtain the biological blood samples necessary for the quantification of the compound tyrphostin AG-17 in concentrations of 10 mg, 3.3 mg and 1 mg in accordance with Good Clinical Practices, always taking care to protect the vulnerability and integrity of the research subjects.

Quantifying the compound tyrphostin AG-17 with a previously validated bioanalytical method.

Estimate the pharmacokinetic parameters of the compound tyrphostin AG-17 at concentrations of 10 mg, 3.3 mg and 1 mg.

Describe the pharmacokinetic parameters of the compound tyrphostin AG-17 in concentrations of 10 mg, 3.3 mg and 1 mg in terms of Cmax, AUC0-t, AUC0-inf and as secondary parameters AUCExt, TMR, Tmax, Ke, t½, Vd and CL and estimate if there are differences by gender.

Establish the possible linearity of the compound tyrphostin AG-17 in concentrations of 10 mg, 3.3 mg and 1 mg.

Correlate the pharmacokinetic markers with the presence of AE or ADRs, with the hemodynamic markers and with the physiological markers and present a dynamic profile of the compound under investigation to propose a pharmacological response that is of potential further interest.

ELIGIBILITY:
Inclusion Criteria:

* Research subjects aged: between 18 and 55 years.
* Sex: 24 men and 24 women.
* Weight: Research subjects with Body Mass Index between 18-27 kg/m2.
* Research subjects with a diagnosis of "HEALTHY"; For this, a clinical history, medical examination, physical examination will be carried out in addition to taking samples to perform clinical analyzes (complete blood count with differential count, to evaluate hematological function, blood chemistry that evaluates pancreatic, renal, hepatic function, cardiac risk, metabolic function, biosafety tests, studies to rule out the presence of hepatitis B and C, HIV and VDRL, general urine test, fasting,). The results of the laboratory tests will be reviewed according to the reference values given by the laboratory and/or the reference values of Instruction I-DCL-VAL-030 "Range of normal values of laboratory tests", the tests The biosafety tests will have to have a NON-REACTIVE result and the cabinet studies (ECG) will have to have a NORMAL diagnosis granted by the Pharmometrica medical staff that evaluates them.
* Research subjects with NEGATIVE results on qualitative drug of abuse tests, breathalyzer and rapid urine pregnancy test (for females), at the beginning of the study.
* Based on the foregoing, the medical staff will determine whether the research subject has the physical capacity to participate in the study. Healthy will be understood as the research subject that meets all the inclusion criteria and does not meet any exclusion criteria.
* Signature of the informed consent for participation in this study, by the IS.

Exclusion Criteria:

* Research subjects with a medical history of allergies.
* Research subjects who have ingested alcoholic beverages, tobacco or xanthines within 48 hours prior to the study.
* Research subjects who have consumed grapefruit, grape, strawberry juice (generally red fruits such as blackberries or blueberries), spicy or charcoal-cooked foods 72 h prior to the study.
* Research subjects who have participated in clinical research studies of any molecule, within 3 months prior to the study date.
* Research subjects who were hospitalized for any reason or were seriously ill within 60 days prior to the study.
* Research subjects who have donated or lost 450 mL or more of blood within 45 days prior to the study.
* Research subjects with disease that require the use of medications Research subjects with medical history of cardiovascular, gastrointestinal, hepatic and/or renal insufficiency.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-07-29 (Estimated)

PRIMARY OUTCOMES:
Tolerance assessment | 30 days
  * Description: type, frequency, duration, consequence, relationship with clinical history, management, follow-up
  * Criteria: severity (serious [serious] and non-serious), severity (mild, moderate and severe)
  * Classification: certain, likely, possible, unlikely, conditional/unclassified, not evaluable/unclassifiable

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmet, S.A de C.V., Mexico City, Azcapotzalco, Mexico

IPD SHARING:
Plan to Share IPD: No
The blood samples obtained as a result of this study will be used to describe a possible change and/or damage in the organism and for the quantification of tyrphostin AG-17, as well as all the data obtained by this research will be evaluated maintaining its confidentiality, adjusting its compliance with the Federal Law on Protection of Personal Data Held by Private Parties